CLINICAL TRIAL: NCT00993421
Title: LY377604 + Sibutramine Hydrochloride Monohydrate: A Phase 2 Weight Loss Efficacy Study in Overweight/Obese Men and Women
Brief Title: A Weight Loss Study in Overweight Men and Women
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical trial terminated due to results from recent nonclinical studies
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11892; I1L-MC-GAEB (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2011-06-02 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — sibutramine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo sibutramine; Drug: Placebo Metoprolol; Drug: Placebo LY377604
- LY377604 (75 mg) (Experimental)
  Interventions: Drug: LY377604; Drug: Placebo sibutramine; Drug: Placebo Metoprolol
- sibutramine (30 mg)/metoprolol (200 mg) (Active Comparator)
  Interventions: Drug: Sibutramine; Drug: Metoprolol
- LY377604 (40 mg)/sibutramine (30 mg) (Experimental)
  Interventions: Drug: LY377604; Drug: Sibutramine; Drug: Placebo Metoprolol
- LY377604 (75 mg)/sibutramine (30 mg) (Experimental)
  Interventions: Drug: LY377604; Drug: Sibutramine; Drug: Placebo Metoprolol
- LY377604 (15 mg)/sibutramine (30 mg) (Experimental)
  Interventions: Drug: LY377604; Drug: Sibutramine; Drug: Placebo Metoprolol
- LY377604 (75 mg)/sibutramine (15 mg) (Experimental)
  Interventions: Drug: LY377604; Drug: Sibutramine; Drug: Placebo Metoprolol

INTERVENTIONS:
Drug: LY377604 — Given daily, orally for 24 weeks
  Arms: LY377604 (15 mg)/sibutramine (30 mg); LY377604 (40 mg)/sibutramine (30 mg); LY377604 (75 mg); LY377604 (75 mg)/sibutramine (15 mg); LY377604 (75 mg)/sibutramine (30 mg)
Drug: Sibutramine — given daily, orally for 24 weeks
  Arms: LY377604 (15 mg)/sibutramine (30 mg); LY377604 (40 mg)/sibutramine (30 mg); LY377604 (75 mg)/sibutramine (15 mg); LY377604 (75 mg)/sibutramine (30 mg); sibutramine (30 mg)/metoprolol (200 mg)
Drug: Metoprolol — given daily, orally for 24 weeks (100 mg for 1 week followed by 200 mg for 23 weeks. Patients unable to tolerate 200 mg will be dose reduced to 100 mg), followed by a 2 week taper (1 week at 100 mg/day followed by 1 week at 50 mg/day).
  Arms: sibutramine (30 mg)/metoprolol (200 mg)
Drug: Placebo sibutramine — given daily, orally for 24 weeks
  Arms: LY377604 (75 mg); placebo
Drug: Placebo Metoprolol — given daily, orally for 26 weeks (24 weeks plus 2 weeks of taper)
  Arms: LY377604 (15 mg)/sibutramine (30 mg); LY377604 (40 mg)/sibutramine (30 mg); LY377604 (75 mg); LY377604 (75 mg)/sibutramine (15 mg); LY377604 (75 mg)/sibutramine (30 mg); placebo
Drug: Placebo LY377604 — given daily, orally for 24 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if LY377604 + sibutramine work better than LY377604 or sibutramine alone in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Are between the body mass index (BMI) of 27 and 45 kg/m^2, inclusive, at the time of screening.

Exclusion Criteria:

* Have a Diastolic Blood Pressure (DBP) greater than 90 mm Hg or less than 55 mm Hg, and/or Systolic Blood Pressure (SBP) >140 mm Hg or <90 mmHg, confirmed by at least 1 repeat measurement. Subjects with hypertension treated with antihypertensive medication are not excluded if blood pressure is within the prescribed limits and they are not treated with excluded medications. Changes in antihypertensive medication are not permitted within 30 days prior to randomization
* Previous history of poorly controlled hypertension, (that is, >160/100 or hypertension which requires more than 2 drugs for control).
* Have a pulse rate >90 bpm or <50 bpm.
* Evidence or history of prior significant cardiovascular disease, coronary artery disease, cardiovascular surgery, significant valvular disease, heart failure, arrhythmias, sick sinus syndrome or stroke.
* Current treatment with β-blockers, calcium channel blockers, digitalis glycosides (for example, digoxin, etc), or clonidine.
* Recent treatment (within 2 weeks prior to randomization) with catecholamine-depleting drugs (such as reserpine or tetrabenazine, monoamine oxidase inhibitors (MAOIs).
* Current treatment with serotonergic drugs, such as selective serotonin reuptake inhibitors (SSRI), any drug that is a serotonin, norepinephrine, or dopamine reuptake inhibitor, "triptan" or ergot therapies for migraine or nausea, or serotonin-releasing agents.
* Treatment with significant inhibitors of Cytochrome P2D6 (CYP2D6), such as bupropion, fluoxetine, paroxetine, quinidine, duloxetine, amiodarone, cimetidine, chlorpheniramine, clomipramine, doxepin, haloperidol, methadone, mibefradil, and ritonavir.
* Participants with bronchospastic diseases or who are treated with bronchodilators or other prescription or nonprescription beta adrenergic agonists.
* Peripheral vascular disease
* History of thyrotoxicosis
* History of seizures (except for childhood febrile convulsion) or at increased risk of seizures (for example, history of significant head trauma or intracranial surgery).
* Have had a significant change in weight, defined as a gain or loss of at least 4 kg (9 lb) in the 90 days prior to randomization
* Have had bariatric surgery (for example, gastric banding or gastric bypass)
* Have had liposuction within 90 days prior to randomization
* Have a disease that affects adipose mass or distribution of energy balance (for example, Cushing's syndrome, uncontrolled hyper- or hypothyroidism).
* Have taken in the 30 days prior to randomization, a medication, herbal product, or nutritional supplement that affects adipose mass or distribution or energy balance, such as glucocorticoids, antiretrovirals, atypical antipsychotics, lithium, valproic acid, lamotrigine, or other anticonvulsants, mirtazapine, bupropion, phentermine, sibutramine, orlistat, rimonabant, amphetamine, or ephedra-containing supplements. Note: Medications that have small and transient effects on weight or medications that may affect weight independent of adipose mass (for example, estrogens or diuretics), may be continued, but may not be started, stopped, or changed during the course of the study.
* Have been diagnosed with an eating disorder, such as anorexia, bulimia, binge eating disorder, or nocturnal eating disorder.
* Have diabetes mellitus treated with medication, or type 2 diabetes mellitus managed with diet and exercise with hemoglobin A1c (HbA1C) >7.0%.
* Symptomatic cholelithiasis in the 90 days prior to randomization.
* Any lifetime history of suicide attempt.
* History of major depressive disorder in the last 2 years or any lifetime history of severe psychiatric disorders (for example, schizophrenia or bipolar disorder).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM-5 PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avon, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomington, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carmel, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sterling Heights, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo LY377604: given orally, daily for 24 weeks.
  Placebo sibutramine: given orally, daily for 24 weeks.
  Placebo metoprolol: given orally, daily for 24 weeks, followed by 2 week taper.
- LY377604 (75 mg): Given orally, daily for 24 weeks.
- Sibutramine (30 mg)/Metoprolol (200 mg): sibutramine (30 mg): Given orally, daily for 24 weeks.
  metoprolol (200 mg): Given orally, daily 100 mg for 1 week followed by 200 mg for 23 weeks (Patients unable to tolerate 200 mg will be dose reduced to 100 mg), followed by a 2 week taper - 1 week at 100 mg/day followed by 1 week at 50 mg/day.
  Placebo LY377604: given orally, daily for 24 weeks.
- LY377604 (15 mg)/Sibutramine (30 mg): LY377604 (15 mg): Given orally, daily for 24 weeks.
  sibutramine (30 mg): Given orally, daily for 24 weeks.
  Placebo metoprolol: Given orally, daily for 24 weeks.
- LY377604 (40 mg)/Sibutramine (30 mg): LY377604 (40 mg): Given orally, daily for 24 weeks.
  sibutramine (30 mg): Given orally, daily for 24 weeks.
  Placebo metoprolol: Given orally, daily for 24 weeks, followed by 2 week taper.
- LY377604 (75 mg)/Sibutramine (30 mg): LY377604 (75 mg): Given orally, daily for 24 weeks.
  sibutramine (30 mg): Given orally, daily for 24 weeks.
  Placebo metoprolol: Given orally, daily for 24 weeks, followed by 2 week taper.
- LY377604 (75 mg)/Sibutramine (15 mg): LY377604 (75 mg): Given orally, daily for 24 weeks.
  sibutramine (15 mg): Given orally, daily for 24 weeks.
  Placebo metoprolol: Given orally, daily for 24 weeks, followed by 2 week taper.
Period: Overall Study
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Started | 49 | 49 | 48 | 49 | 52 | 50 | 46
Completed | 5 | 4 | 5 | 4 | 6 | 4 | 4
Not Completed | 44 | 45 | 43 | 45 | 46 | 46 | 42
Not completed — Adverse Event | 2 | 7 | 6 | 9 | 5 | 7 | 1
Not completed — Sponsor Decision | 36 | 31 | 28 | 30 | 38 | 30 | 29
Not completed — Lost to Follow-up | 3 | 5 | 5 | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 3 | 2 | 3 | 3 | 3 | 5 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Entry Criteria Exclusion | 0 | 0 | 1 | 3 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg) | Total
Number analyzed (Participants) | 49 | 49 | 48 | 49 | 52 | 50 | 46 | 343
Age Continuous [Mean (Standard Deviation); unit: years] | 42.71 (10.86) | 43.89 (11.02) | 44.68 (12.00) | 43.42 (11.06) | 44.15 (10.71) | 45.80 (9.15) | 43.93 (10.15) | 44.09 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 38 | 39 | 40 | 41 | 34 | 275
  Male | 8 | 7 | 10 | 10 | 12 | 9 | 12 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Black or African American | 12 | 5 | 8 | 10 | 8 | 6 | 7 | 56
  White | 36 | 43 | 39 | 34 | 43 | 42 | 36 | 273
  More than one race | 1 | 1 | 1 | 3 | 1 | 1 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 48 | 49 | 52 | 50 | 46 | 343
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 166.10 (8.02) | 166.86 (8.40) | 167.51 (9.22) | 165.23 (8.93) | 168.13 (7.88) | 168.99 (8.18) | 168.38 (7.50) | 167.32 (8.34)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 97.92 (18.73) | 97.15 (15.67) | 102.25 (17.80) | 96.36 (18.08) | 99.09 (17.73) | 100.96 (17.20) | 100.09 (17.11) | 99.10 (17.46)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight (kilograms) divided by height (meters) squared.
  kilograms/square meters (kg/m^2) | 35.22 (4.96) | 34.78 (4.53) | 36.34 (5.36) | 35.12 (4.55) | 34.86 (4.39) | 35.30 (4.44) | 35.22 (4.87) | 35.26 (4.71)
Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic Blood Pressure (SBP) | 117.11 (11.53) | 115.72 (10.78) | 117.35 (10.13) | 118.67 (11.11) | 118.34 (11.37) | 119.86 (11.42) | 120.72 (11.36) | 118.24 (11.13)
  Diastolic Blood Pressure (DBP) | 75.12 (7.31) | 74.40 (7.70) | 75.83 (6.76) | 76.61 (7.07) | 76.94 (6.31) | 77.87 (6.82) | 78.38 (6.23) | 76.44 (6.97)
Waist and Hip Circumference [Mean (Standard Deviation); unit: centimeters (cm)]
  Waist Circumference | 109.13 (14.10) | 107.42 (10.70) | 111.47 (12.58) | 107.31 (12.06) | 110.18 (10.80) | 109.99 (11.49) | 109.15 (12.95) | 109.24 (12.10)
  Hip Circumference | 119.76 (12.36) | 118.55 (9.42) | 120.29 (11.51) | 117.65 (11.13) | 117.30 (14.96) | 119.43 (11.45) | 118.01 (11.43) | 118.70 (11.83)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight From Baseline to 24 Week Endpoint
Description: Body weight percentage change from baseline is presented as Least Squares Mean (LSMean) with treatment, visit, and their interaction as fixed effects, subject as a random effect, baseline body weight, age, gender were used as covariates.
Time Frame: Baseline, 24 weeks
Population: ITT population: all randomized participants receiving at least 1 dose of the study drug according to the treatment the participants actually received. Participants with baseline and a measurement at endpoint were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 28 | 26 | 24 | 25 | 32 | 22 | 23
percent change | -2.21 (0.81) | 0.48 (0.84) | -6.12 (0.86) | -8.53 (0.80) | -6.61 (0.79) | -7.05 (0.85) | -4.71 (0.86)
Statistical Analysis 1: Comparison: LY377604 (75 mg) vs LY377604 (15 mg)/Sibutramine (30 mg); Hypothesis: Treatment with a combination of LY377604 + sibutramine for 24 weeks would result in weight loss that was significantly greater than treatment with either sibutramine or LY377604 alone; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: LY377604 (75 mg) vs LY377604 (40 mg)/Sibutramine (30 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: LY377604 (75 mg) vs LY377604 (75 mg)/Sibutramine (30 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 4: Comparison: LY377604 (75 mg) vs LY377604 (75 mg)/Sibutramine (15 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 5: Comparison: Sibutramine (30 mg)/Metoprolol (200 mg) vs LY377604 (15 mg)/Sibutramine (30 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.041, Mixed Models Analysis
Statistical Analysis 6: Comparison: Sibutramine (30 mg)/Metoprolol (200 mg) vs LY377604 (40 mg)/Sibutramine (30 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis
Statistical Analysis 7: Comparison: Sibutramine (30 mg)/Metoprolol (200 mg) vs LY377604 (75 mg)/Sibutramine (30 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.437, Mixed Models Analysis
Statistical Analysis 8: Comparison: Sibutramine (30 mg)/Metoprolol (200 mg) vs LY377604 (75 mg)/Sibutramine (15 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.249, Mixed Models Analysis

2. Secondary Outcome: The Mean Change in Body Weight From Baseline to 24 Week Endpoint
Description: Body weight change from baseline is presented as Least Squares Mean (LSMean) with treatment, visit, and their interaction as fixed effects, subject as a random effect, baseline body weight, age, gender were used as covariates.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 28 | 26 | 24 | 25 | 32 | 22 | 23
kilograms | -2.37 (0.82) | 0.45 (0.85) | -6.41 (0.87) | -8.15 (0.81) | -6.49 (0.79) | -7.06 (0.85) | -4.68 (0.87)

3. Secondary Outcome: Percentage of Participants Who Achieve a Minimum of 10% Weight Loss From Baseline at 24 Weeks
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 49 | 49 | 48 | 49 | 52 | 50 | 46
percentage of participants | 10.2 | 0.0 | 18.8 | 34.7 | 21.2 | 18.0 | 6.5

4. Secondary Outcome: Change in Heart Rate From Baseline to 24 Week Endpoint
Description: Heart rate change from baseline is presented as Least Squares Mean (LSMean) with treatment, visit, and their interaction as fixed effects, subject as a random effect, baseline heart rate, age, gender were used as covariates.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 30 | 27 | 24 | 26 | 33 | 22 | 25
beats per minute (bpm) | -0.69 (1.51) | -3.34 (1.60) | -1.37 (1.67) | 6.11 (1.60) | 2.19 (1.44) | -2.66 (1.72) | -2.46 (1.63)

5. Secondary Outcome: Change in Blood Pressure From Baseline to 24 Week Endpoint
Description: Blood pressure change from baseline is presented as Least Squares Mean (LSMean) with treatment, visit, and their interaction as fixed effects, subject as a random effect, baseline blood pressure, age, gender were used as covariates.
Time Frame: Baseline, 24 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 30 | 27 | 24 | 26 | 33 | 22 | 25
mm Hg
  Systolic Blood Pressure | -2.84 (1.67) | -3.59 (1.75) | -3.77 (1.84) | 3.25 (1.76) | -1.17 (1.59) | -0.43 (1.90) | 0.95 (1.80)
  Diastolic Blood Pressure | -2.25 (1.28) | -3.84 (1.35) | -2.51 (1.41) | 2.03 (1.34) | 0.13 (1.22) | -2.87 (1.45) | -0.38 (1.38)

6. Secondary Outcome: Change in Body Composition Using Dual Energy X-ray Absorptiometry (DXA) From Baseline to 24 Week Endpoint
Description: Change in body composition (lean body mass and fat mass) was assessed using dual energy x-ray absorptiometry (DXA) and is presented as LSMEAN values with treatment, visit, and their interaction as fixed effects, subject as a random effect, baseline body composition, age, gender were used as covariates.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 28 | 23 | 23 | 23 | 31 | 21 | 25
kilograms (kg)
  Fat Mass | -2.40 (0.72) | 0.54 (0.76) | -3.00 (0.75) | -6.13 (0.71) | -4.80 (0.67) | -4.29 (0.77) | -2.55 (0.73)
  Lean Mass | -0.55 (0.41) | 0.15 (0.45) | -1.92 (0.45) | -1.85 (0.43) | -0.71 (0.39) | -1.08 (0.47) | -1.48 (0.43)

7. Secondary Outcome: Change in Waist Circumference From Baseline to 24 Week Endpoint
Description: Change from baseline to endpoint is presented as LSMEAN with treatment, visit, and their interaction as fixed effects, subject as a random effect, baseline waist circumference, age, gender were used as covariates.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: centimeter (cm)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 31 | 27 | 24 | 25 | 32 | 22 | 25
centimeter (cm) | -6.58 (2.44) | -2.51 (2.62) | -8.84 (2.77) | -6.76 (2.71) | -3.57 (2.38) | -3.55 (2.88) | -8.67 (2.68)

8. Secondary Outcome: Percentage Change in Waist Circumference From Baseline to 24 Week Endpoint
Description: Percentage change from baseline to endpoint is presented as LSMEAN with treatment, visit, and their interaction as fixed effects, subject as a random effect, baseline waist circumference, age, gender were used as covariates.
Time Frame: Baseline, 24 weeks
Population: ITT
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 31 | 27 | 24 | 25 | 32 | 22 | 25
percent change | -5.86 (2.21) | -2.22 (2.38) | -7.55 (2.52) | -5.96 (2.46) | -3.02 (2.16) | -3.11 (2.62) | -7.29 (2.44)

9. Secondary Outcome: Change in Total Cholesterol From Baseline to 24 Weeks Endpoint
Time Frame: Baseline, 24 weeks
Population: Intent to Treat (IIT) population: all randomized participants who received at least one dose of study drug and received the intended study drug. Participants with baseline and at least one post-baseline measurement were included in the analysis (LOCF).
Measure: Mean (Standard Deviation); unit: millimole/Liter (mmol/L)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 48 | 49 | 45 | 49 | 48 | 50 | 43
millimole/Liter (mmol/L) | -0.12 (0.68) | -0.13 (0.47) | -0.04 (0.69) | -0.01 (0.67) | 0.00 (0.68) | 0.17 (0.70) | -0.13 (0.76)

10. Secondary Outcome: Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to 24 Weeks Endpoint
Time Frame: Baseline, 24 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole/Liter (mmol/L)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 48 | 49 | 45 | 49 | 48 | 50 | 43
millimole/Liter (mmol/L) | -0.02 (0.16) | -0.05 (0.19) | -0.03 (0.15) | 0.01 (0.15) | 0.06 (0.21) | 0.01 (0.17) | -0.04 (0.17)

11. Secondary Outcome: Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to 24 Weeks Endpoint
Time Frame: Baseline, 24 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole/Liter (mmol/L)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 48 | 49 | 45 | 49 | 48 | 49 | 43
millimole/Liter (mmol/L) | -0.07 (0.57) | -0.03 (0.44) | 0.00 (0.62) | -0.00 (0.58) | -0.07 (0.50) | 0.16 (0.65) | -0.16 (0.67)

12. Secondary Outcome: Change in Triglycerides From Baseline to 24 Weeks Endpoint
Time Frame: Baseline, 24 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millimole/Liter (mmol/L)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 48 | 49 | 45 | 49 | 48 | 50 | 43
millimole/Liter (mmol/L) | -0.06 (0.61) | -0.11 (0.48) | -0.04 (0.66) | 0.04 (0.60) | 0.04 (0.55) | 0.03 (0.72) | 0.22 (0.94)

13. Secondary Outcome: Change From Baseline for Obesity Weight Loss Quality of Life Instrument (OWL-QoL)
Description: Results presented as Least Squares Mean with treatment, visit, and their interaction as fixed effects, subject as random effect, baseline body mass index used as covariate. OWL-QoL consists of 17 items on scale ranging from 0 (Not at all) to 6 (A very great deal). Before calculating scores, each item is reversed. A single quality of life score is computed by summing each item and transforming this raw score onto standardized scale of 0 (greatest impact) to 100 (lowest impact) using formula: score = [(sum of component items score (minus) lowest possible score/ possible raw score range)*100].
Time Frame: Baseline, 24 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 31 | 26 | 24 | 26 | 34 | 23 | 26
units on a scale | 11.71 (4.93) | 2.67 (5.30) | 13.96 (5.26) | 16.52 (5.27) | 17.44 (5.17) | 13.53 (5.35) | 14.02 (5.23)

14. Secondary Outcome: Change From Baseline in Vitality Scale of Medical Outcomes Short Form - 36 (SF-36) Scale
Description: Vitality change from baseline is presented as Least Squares Mean (LSMean) with treatment, visit, and their interaction as fixed effects, subject as a random effect, baseline body mass index was used as covariate. SF-36 is a self-reported questionnaire that consists of 36 questions covering 8 health domains including vitality. The vitality domain results are presented. The vitality domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning.
Time Frame: Baseline, 24 weeks
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 31 | 27 | 24 | 25 | 34 | 24 | 26
units on a scale | 10.79 (5.24) | 5.83 (5.66) | 16.81 (5.63) | 10.69 (5.69) | 7.35 (5.53) | 10.62 (5.72) | 13.61 (5.58)

15. Secondary Outcome: Change in Glycated Hemoglobin A1c (HbA1c) From Baseline
Description: Analysis of change in HbA1c was not conducted due to an inadequate number of samples.
Time Frame: Baseline, 24 weeks
Population: Zero participants were analyzed due to the small sample size.
Measure: Mean (Standard Deviation); unit: percent glycated hemoglobin
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Change in Fasting Glucose From Baseline to 24 Weeks Endpoint
Description: Analysis of change in fasting glucose was not conducted due to an inadequate number of samples.
Time Frame: Baseline, 24 weeks
Population: Zero participants were analyzed due to an inadequate number of samples.
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Change in Fasting Insulin From Baseline to 24 Weeks Endpoint
Description: Analysis of change in fasting insulin was not conducted due to an inadequate number of samples.
Time Frame: Baseline, 24 weeks
Population: Zero participants were analyzed due to an inadequate number of samples.
Measure: Mean (Standard Deviation); unit: micro Units/milliliter (μU/mL)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Change in Insulin Resistance From Baseline to 24 Weeks Endpoint
Description: Analysis of change in insulin resistance was not conducted due to an inadequate number of samples.
Time Frame: Baseline, 24 weeks
Population: Zero participants were analyzed due to inadequate number of samples.
Measure: Mean (Standard Deviation); unit: Units of Insulin/Day
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve (AUC)
Description: Analysis of AUC was not conducted due to an inadequate number of samples collected.
Time Frame: 4 weeks, 12 weeks, and 24 weeks
Population: Zero participants were analyzed because of the low sample size.
Measure: Geometric Mean (Standard Error); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax)
Description: Analysis of Cmax was not conducted due to an inadequate number of samples collected.
Time Frame: 4 weeks, 12 weeks, and 24 weeks
Population: Zero participants were analyzed due to the small sample size.
Measure: Geometric Mean (Standard Error); unit: nanograms per milliliter (ng/mL)
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30 mg)/Metoprolol (200 mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Sibutramine (30mg)/Metoprolol (200mg): sibutramine (30 mg): Given orally, daily for 24 weeks.
  metoprolol (200 mg): Given orally, daily 100 mg for 1 week followed by 200 mg for 23 weeks (Patients unable to tolerate 200 mg will be dose reduced to 100 mg), followed by 2 week taper (1 week at 100 mg/day followed by 1 week at 50 mg/day).
  Placebo LY377604: given orally, daily for 24 weeks.
- LY377604 (15 mg)/Sibutramine (30 mg): LY377604 (15 mg): Given orally, daily for 24 weeks.
  sibutramine (30 mg): Given orally, daily for 24 weeks.
  Placebo metoprolol: Given orally, daily for 24 weeks, followed by 2 week taper.
Arm/Group | Placebo | LY377604 (75 mg) | Sibutramine (30mg)/Metoprolol (200mg) | LY377604 (15 mg)/Sibutramine (30 mg) | LY377604 (40 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (30 mg) | LY377604 (75 mg)/Sibutramine (15 mg)
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 2/48 | 2/49 | 0/52 | 1/50 | 2/46
Other Adverse Events (participants affected / at risk) | 41/49 | 39/49 | 38/48 | 44/49 | 43/52 | 46/50 | 33/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | LY377604 (75 mg) (N=49) | Sibutramine (30mg)/Metoprolol (200mg) (N=48) | LY377604 (15 mg)/Sibutramine (30 mg) (N=49) | LY377604 (40 mg)/Sibutramine (30 mg) (N=52) | LY377604 (75 mg)/Sibutramine (30 mg) (N=50) | LY377604 (75 mg)/Sibutramine (15 mg) (N=46)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — This event (result of automobile accident) resulted in death.
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | LY377604 (75 mg) (N=49) | Sibutramine (30mg)/Metoprolol (200mg) (N=48) | LY377604 (15 mg)/Sibutramine (30 mg) (N=49) | LY377604 (40 mg)/Sibutramine (30 mg) (N=52) | LY377604 (75 mg)/Sibutramine (30 mg) (N=50) | LY377604 (75 mg)/Sibutramine (15 mg) (N=46)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 11 (11) | 9 (9) | 7 (8) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 5 (6) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 4 (4) | 6 (6) | 20 (20) | 16 (16) | 10 (12) | 8 (9)
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0) | 3 (3) | 4 (5) | 2 (2) | 3 (3) | 2 (4)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 5 (5) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Sinusitis (Infections and infestations) | 2 (3) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 6 (9) | 4 (4) | 2 (2) | 4 (4) | 4 (4) | 5 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 4 (4) | 4 (4)
Viral infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 5 (6) | 2 (3) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 1 (1) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 4 (4) | 4 (4) | 7 (8) | 6 (6) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 5 (5) | 5 (5) | 5 (6) | 4 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (3) | 3 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (5) | 3 (3) | 8 (8) | 7 (7) | 6 (6) | 2 (2)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (4) | 2 (2) | 1 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days